CLINICAL TRIAL: NCT04929730
Title: Effect of Organisation of Medical Care on Health Status in Patients With Acute Kidney Injury
Brief Title: Effect of Medical Care on Health Status in Acute Kidney Injury
Acronym: EMESA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medizinisches Versorgungszentrum Diaverum Potsdam (Other)
Collaborators: Ernst von Bergmann Hospital (Other); University of Magdeburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1.1
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Acute Renal Insufficiency
Keywords: Nephrologists; Health Services, Outpatient; Patient Care Bundles
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: alternating cluster-randomised allocation of investigation-periods alternierende Cluster-randomisierte Zuordnung der Untersuchungszeiträume
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients with an acute kidney injury in laborytory testing receive usual care. Nephrology co-supervision only on enquiry of the ward physician
- Interventional group (Other): Patients with an acute kidney injury in laborytory testing receive nephrology co-supervision in hospital and information about the importance of ambulant follow-up care.
  Interventions: Other: Nephrology care bundle

INTERVENTIONS:
Other: Nephrology care bundle — Nephrology care bundle
  Arms: Interventional group

SUMMARY:
Various forms of organisation in the care of patients with akute kidney injury are investigated.

In this prospective study the investigators compare the effect of usual care with the effect of intensive care. Primary endpoint is the development of cardiovascular events ("major adverse cardiovascular events" "MACE").

DETAILED DESCRIPTION:
The investigators plan to investigate the use of various organisation forms in the care of patients with the diagnosis of acute kidney injury in the hospital. This prospective study compares the effect of usual care with the effect of intensive care in the hospital and outpatient health care center. Primary endpoint is the development of cardiovascular events ("major adverse cardiovascular events" "MACE"). Patients with intensive care receive a nephrology consulting report and extensive information about acute kidney injury and the importance of ambulant follow-up care.

The investigators hypothesise a better in-hospital treatment and an improvement of clinical course in the interventional group.

ELIGIBILITY:
Inclusion Criteria:

* men and women at the age of 18 or older
* acute kidney injury according to KDIGO-guidelines
* The patient (or his/ her authorised representative) is in the position and willing to give informed consent.

Exclusion Criteria:

* Patients, who received kidney transplantation
* Patients on chronic dialysis at the time of enrolment
* Patients who are placed in an institution by judicial or governmental order
* Pregnancy
* Infection with HI- or Infektionen mit HI- oder Hepatitis virus infektion
* Participation in a clinical study with testing on drugs or medical devices (according to German Medicines Law or Medicinal Devices Act)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 months
  major adverse cardiovascular event

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haase, Prof, Principal Investigator — Medizinische Fakultät d. Otto-v-Guericke-Universität Magdeburg, MVZ Diaverum Am Neuen Garten Potsdam
Locations (1):
- Ernst von Bergmann Hospital, Potsdam, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haase M, Kribben A, Zidek W, Floege J, Albert C, Isermann B, Robra BP, Haase-Fielitz A. Electronic Alerts for Acute Kidney Injury. Dtsch Arztebl Int. 2017 Jan 9;114(1-02):1-8. doi: 10.3238/arztebl.2017.0001. PMID 28143633
- [Background] Holmes J, Rainer T, Geen J, Roberts G, May K, Wilson N, Williams JD, Phillips AO; Welsh AKI Steering Group. Acute Kidney Injury in the Era of the AKI E-Alert. Clin J Am Soc Nephrol. 2016 Dec 7;11(12):2123-2131. doi: 10.2215/CJN.05170516. Epub 2016 Oct 28. PMID 27793961
- [Background] Lachance P, Villeneuve PM, Rewa OG, Wilson FP, Selby NM, Featherstone RM, Bagshaw SM. Association between e-alert implementation for detection of acute kidney injury and outcomes: a systematic review. Nephrol Dial Transplant. 2017 Feb 1;32(2):265-272. doi: 10.1093/ndt/gfw424. PMID 28088774
- [Background] Chawla LS, Amdur RL, Shaw AD, Faselis C, Palant CE, Kimmel PL. Association between AKI and long-term renal and cardiovascular outcomes in United States veterans. Clin J Am Soc Nephrol. 2014 Mar;9(3):448-56. doi: 10.2215/CJN.02440213. Epub 2013 Dec 5. PMID 24311708